CLINICAL TRIAL: NCT05036577
Title: A Dose-escalating Pilot Study of Orelabrutinib in Combination With Rituximab, Methotrexate and Dexamethasone for Newly-diagnosed Primary Central Nervous System Lymphoma
Brief Title: A Dose-escalating Pilot Study of Orelabrutinib for Newly-diagnosed PCNSL
Acronym: ORMD2021
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Tong Chen, MD, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-726
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — orelabrutinib; Rituximab; Methotrexate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ORMD (Orelabrutinib, Rituximab, Methotrexate and Dexamethasone) (Experimental): Patients were treated for 6-8 cycles of induction therapy with 21 days per cycle, receiving rituximab (375mg/m2 on day 1), dexamethasone (10-15mg on d1-d4), MTX (d2, 3.5g/m2 or 5g/m2), and orelabrutinib (once daily, after MTX clearance, 150mg/d, or 200mg/d), followed by orelabrutinib maintenance up to one year among CR/CRu patients or until disease progression, intolerable toxicity, death, informed consent withdrawal or lost of follow up (whichever occurs first). The primary objective was to determine the maximum tolerated dose (MTD) of the combination of orelabrutinib and MTX with R and D and investigate the safety and tolerability of this regimen using Bayesian Optimal Interval (BOIN) waterfall design to determine rule of dose escalation and movement among dose combination matrix to identify MTD contour.
  Interventions: Drug: Orelabrutinib; Drug: Rituximab; Drug: Methotrexate (MTX); Drug: Dexamethasone

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib will be given as 150 mg/d or 200 mg/d orally 72h after MTX infusion or MTX clearance, every 21 days for 6-8 cycles during combination induction treatment.
  Daily Orelabrutinb with dose in last cycle of induction will be administered as maintenance treatment for up to 1 year or until disease progression, intolerable toxicity, death, informed consent withdrawal or lost of follow up (whichever occurs first).
Drug: Rituximab — Rituximab 375 mg/m2 intravenous infusion d1, every 21 days for 6-8 cycles during combination induction treatment.
Drug: Methotrexate (MTX) — high-dose Methotrexate 3.5 g/m2 or 5g/m2 intravenous infusion (3h) d2, every 21 days for 6-8 cycels during combination induction treatment.
Drug: Dexamethasone — Dexamethasone 10-15 mg, iv, d1-4, every 21 days for 6-8 cycles during combination induction treatment.

SUMMARY:
This is a single arm, single center, open label pilot study of Orelabrutinib combined with Rituximab, high-dose (HD) Methotrexate and Dexamethasone in newly-diagnosed primary central nervous system lymphpoma (PCNSL). The purpose is to evaluate the safety and to find the optimal dose of Orelabrutinib and Methotrexate in this combination treatment for newly-diagnosed PCNSL patients.

DETAILED DESCRIPTION:
The eligible patients will be treated with Orelabrutinib combined with Rituximab, high-dose Methotrexate and Dexamethasone during induction treatment (6-8 cycles; 21 days/cycle): Rituximab 375 mg/m2, intravenous infusion, d1; HD-MTX 3.5 g/m2 intravenous infusion (3h), d2; Dexamethasone 10-15 mg, iv, d1-4. Orelabrutinib will be given 72h after MTX infusion or until MTX clearance. The study will investigate optimal dose combination of Orelabrutinib and MTX implementing BOIN waterfall design. The starting dose of Orelabrutinib is 150 mg/d and the dose will be escalated to 200 mg/d, throughout the whole cycle. Meanwhile, the starting dose of MTX is 3g/m2 and will be escalated to 5g/m2, throughout induction phase. Dose escalation and movement in dose matrix will be determined by BOIN algorithm. For CR/CRu patients after completion of induction treatment, daily Orelabrutinib will be administered as maintenance treatment for up to 1 year or until disease progression, intolerable toxicity, death, informed consent withdrawal or lost of follow up (whichever occurs first). Patients will be evaluated every 2 cycles during induction therapy and every 12 weeks during maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* anti-neoplasm systemic treatement naive primary central nervous system lymphoma
* Pathological type is diffuse large B cell lymphoma
* Enough residual sample of tumor after pathological diagnosis
* ECOG =<3
* Life expectancy >3 months
* Adequate organ function and adequate bone marrow reserve
* Must be able to tolerate lumbar puncture and/or have Omaya tube
* Participant or his/her legal agent must be willing to sign a written informed consent document.

Exclusion Criteria:

* Lymphoma invading outside CNS
* Lymphoma only existed in vitreo-retina
* Severe or uncontrolled cardiovascular disease
* Active hemorrhage within 2 months prior screening
* Cerebral ischemic stroke or bleeding within 6 months prior screening
* Organ transplantation or allogeneic hematopoietic stem cell transplantation history
* Other surgery history within 6 weeks prior screening
* Anti-tumor herbal medicine treatment within 4 weeks prior screening
* Activated or uncontrolled hepatitis virus B infection (HBsAg positive with/or HBc Ab positive and HBV-DNA titration positive), hepatitis virus C antibody positive, HIV positive.
* Uncontrolled active systemic fungal, bacterial, virus or other microbe infection, or intravenous injection of antibiotics needed
* Accepted live vaccine or immunization within 4 weeks prior eligibility
* Continuously taking drugs with medium / strong inhibition or induction of cytochrome P450 CYP3A is needed
* Allergy to orelabrutinib or the subsidiary (or supplementary) material (Hydroxypropyl methylcellulose acetate succinate, mannitol, cross-linked sodium carboxymethylcellulose, hydroxypropyl cellulose, silica and magnesium stearate)
* Obvious gastro-bowel disease which may influence the intaking, transportation or absorption of the drug, or total gastrectomy
* Past or present pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, or drug-related pneumonia, with severe impairment of pulmonary function
* Chronic liver damage, severe fatty liver or alcoholic liver disease
* Intention to undergo autologous stem cell transplantation
* Pregnant or breeding women, or women of childbearing age who are unwilling to take contraceptive measures during the whole study period and within 180 days after the last administration of the study drug; non surgically sterilized men who are unwilling to take contraceptive measures during the whole study period and within 180 days of the last administration of the study drug.
* Potentially life-threatening situation, or severe organ dysfunction, or situations the researchers believe not suitable for the trial
* Any mental or cognitive impairment which may limit the understanding and implementation of informed consent or the compliance with the study.
* previously exposed with WBRT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
define the Maximum tolerated dose (MTD) contour of Orelabrutinib and MTX | From the start of the first dose of Orelabrutinib to the end of the first cycle of induction treatment (21 days/cycle)
  A BOIN waterfall design will be employed. Two dose levels of Orelabrutinib (dose level 1: 150 mg/d, dose level 2: 200 mg/d) and two dose levels of MTX (dose level 1: 3.5g/m2, dose level 2: 5g/m2) will be investigated, generating 4 dose combination. DLT was defined by the occurrence of severe toxicities during the first cycle: any grade 4 hematologic toxicity, grade 3 febrile neutropenia and grade 3 thrombocytopenia with hemorrhage, or any grade 3 non-hematologic toxicity that failed to respond to supportive therapy and possibly related to orelabrutinib and/or MTX (assessed according to NCI CTCAE V5.0)

SECONDARY OUTCOMES:
ORRi | At the end of cycle 6-8 (each cycle is 21 days)
  ORRi is defined as the proportion of patients with a best response of CR, CRu or PR during induction therapy
CRi | At the end of cycle 6-8 (each cycle is 21 days)
  CRi is defined as the proportion of patients with a best response of CR or CRu during induction treatment
TTR | At the end of cycle 6-8 (each cycle is 21 days)
  Time to response during induction therapy
ORRm | At the end of completion of 1 year of maintenance treatment
  ORRm is defined as the proportion of patients with a best response of CR, CRu or PR during maintenance therapy
CRm | At the end of completion of 1 year of maintenance treatment
  CRm is defined as the proportion of patients with a best response of CR or CRu during maintenance therapy
Progression-free survival | Up to 2 years
  Progression-free survival is calculated from the date of start of therapy until the date of first documented progress or death due to any cause.
Overall survival | Up to 2 years
  Overall survival is defined as the duration from start of treatment to time of death.

OTHER OUTCOMES:
concentration of Orelabrutinib | The blood and CSF concentration of Orelabrutinib will be evaluated 1.5-2 hours after Orelabrutinib administration before first day of cycle 3.(each cycle is 21 days)
  To detect the blood and CSF concentration of Orelabrutinib
gene mutations and frequency | At baseline
  The types of gene mutations and frequency of tumor are measured by whole exon sequencing.
cytokine in the CSF | At the baseline, day 1 at cycle 3, 5 (21 days/cycle), and every 3 months in the maintenance stage (up to 1 year))
  The levels of cytokine will be analyzed by flow cytometry.
circulating tumor DNA (ctDNA) in the CSF | At the baseline, day 1 at cycle 3, 5 (21 days/cycle), and every 3 months in the maintenance stage (up to 1 year))
  The levels of ctDNA will be analyzed by next-generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Tong Chen, Principal Investigator — Huashan Hospital
Locations (1):
- Department of Hematology, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No